CLINICAL TRIAL: NCT05443542
Title: Virtual Reality in Cognitive Rehabilitation of Processing Speed for Persons With Acquired Brain Injury
Brief Title: VIrtual Reality in Cognitive Rehabilitation of Processing Speed for Persons With ABI
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Sunnaas Rehabilitation Hospital (Other)
Collaborators: Oslo Metropolitan University (Other); Norwegian University of Science and Technology (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: VR i kogn rehab av tempo
Record Dates: First submitted 2022-05-19; First posted 2022-07-05 (Actual); Last update posted 2022-11-08 (Actual); Status verified 2022-11

CONDITIONS: Traumatic Brain Injury; Stroke; Acquired Brain Injury; Brain Injuries; Brain Diseases
Keywords: TBI; Traumatic brain injury; Stroke; Acquired brain injury; Virtual Reality; VR; Cognitive rehabilitation
MeSH Terms: conditions — Brain Injuries, Traumatic; Stroke; Brain Injuries; Brain Diseases

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Virtual Reality Group (Experimental): Group 1 will play a VR game using an Oculus Quest 2 in a home setting
  Interventions: Device: Virtual Reality
- Active control group (Active Comparator): The control group will be given a pamphlet containing exercises affecting working memory, attention and processing speed to be performed in a home setting
  Interventions: Other: Control intervention

INTERVENTIONS:
Device: Virtual Reality — Game to be played is a commercially available VR game
  Other Names: Oculus Quest 2
  Arms: Virtual Reality Group
Other: Control intervention — Sodoku, crossword puzzles
  Arms: Active control group

SUMMARY:
One hundred participants with acquired brain injury (ABI) will be included in a randomized controlled trial, with one group playing a commercially available VR game and the control group doing activities in their everyday as cognitive training. The trial aims to investigate how VR can affect processing speed in the ABI population, and if these effects can transfer into everyday activities. The training will be performed in the participants homes, with assistance provided by the project group via phone or video conference. The training period will last five weeks. Participant's cognitive functions will be measured with questionnaires and neuropsychological tests at the start of the training period, at the end of training and sixteen weeks after the start of the intervention. In depth experiences with VR as a training method will be gathered through performing focus group interviews with some of the participants from the VR group, in addition to self-reported questionnaires from all the participants.

DETAILED DESCRIPTION:
A randomized controlled trial (RCT) will be conducted where the experimental intervention is playing a commercial VR game. The VR group will follow a training regime of a 30 min VR session five times per week for 5 weeks. The control group will carry on with treatment as usual, in addition, participants will receive an information booklet covering cognitive training in everyday life. Baseline and outcome measures in terms of neuropsychological assessment and questionnaires will be performed at baseline (T1), at the end of the intervention period (T2) and at the 16-week follow-up (T3).

The VR group will train with a rhythm VR game that is considered as a good candidate for basic training of the multifaceted aspects of attention including speed of information processing, selection, sustained attention, shifting/dividing of attention, and working memory.

The VR game is selected on the grounds of clinical experience with VR training of processing speed, attention and working memory, and is also suggested in research as suitable games for cognitive rehabilitation.

ELIGIBILITY:
Inclusion Criteria:

* Patients in stable phase after Acquired brain injury, minimum one year after injury
* Physically able to operate VR-technology
* Norwegian or English skills adequate to understand instructions, play the VR-games and to provide valid responses to assessment methods

Exclusion Criteria:

* Severe aphasia affecting their understanding of instructions
* Apraxia affecting their ability to use VR-equipment
* Visual neglect
* Severe mental illness, substance abuse or co-existing neurological disorders

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 100 (Estimated)
Dates: Start 2022-09-15 (Actual); Primary Completion 2023-12 (Estimated); Study Completion 2024-12 (Estimated)

PRIMARY OUTCOMES:
Change in processing speed | Measured at baseline, after the intervention period (5 weeks) and at follow-up (16 weeks after baseline)
  Connors Continous Performance test 3rd edition, Coefficient of Variation

SECONDARY OUTCOMES:
Change in patient reported executive functioning | Measured at baseline, after the intervention period (5 weeks) and at follow-up (16 weeks after baseline)
  Behavior Rating Inventory of Executive function (BRIEF-A)
Transfer effect to everyday activities | Measured at baseline, after the intervention period (5 weeks) and at follow-up (16 weeks after baseline)
  Patient Competency Rating Scale
Change in working memory | Measured at baseline, after the intervention period (5 weeks) and at follow-up (16 weeks after baseline)
  Wechslers Adult Intelligence Scale IV, Backwards Digit Span
Change in working memory | Measured at baseline, after the intervention period (5 weeks) and at follow-up (16 weeks after baseline)
  Wechslers Adult Intelligence Scale IV, Digit sequencing test
Change in informant reported executive functioning | Measured at baseline, after the intervention period (5 weeks) and at follow-up (16 weeks after baseline)
  Behavior Rating Inventory of Executive function (BRIEF-A)
Change in sustained attention | Measured at baseline, after the intervention period (5 weeks) and at follow-up (16 weeks after baseline)
  Connors Continous Performance test 3rd edition, Performance variability over time

CONTACTS AND LOCATIONS:
Overall Officials: Marianne Løvstad, PhD, Principal Investigator — Sunnaas Rehabilitation hopsital
Locations (1):
- Sunnaas Rehabilitation Hospital, Nesoddtangen, Akershus, Norway

IPD SHARING:
Plan to Share IPD: No
Data will be deidentified and will not be made publicly available due to data protection regulations